CLINICAL TRIAL: NCT06713161
Title: Tumor-Targeted-NIR-II Fluorescent Molecular Probes for the Identification of Breast Cancer Tissue and SLN Metastatic Status
Acronym: NIR-II
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Xiang'an Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2024-240
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Metastases; Margin Assessment
Keywords: NIR-II; Breast Cancer; Sentinel Lymph Node; Surgical Navigation; Metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NIR-II probe incubation: The fresh excision breast tissues or SLN will be completely soaked in the NIR-II probe (i.e:ICG-POL6326) incubation solution (12.5,25,50,100 ug/mL) for1, 3, 5,7 or 10 min, followed by 5 min of rinsing with PBST buffer and drying with absorbent paper.The NIR-II fluorescence imaging will be then performed under the DPM NIR-II system. And the correlation between pathological characterization and fluorescent information will be further analyzed.
  Interventions: Diagnostic Test: NIR-II Probe(i.e ICG-POL6326) incubation solution

INTERVENTIONS:
Diagnostic Test: NIR-II Probe(i.e ICG-POL6326) incubation solution — After the tissues were incubated with the optimal concentration of the NIR-II probe for the appropriate time, the tissues were washed with the eluate, and then the fluorescence intensity of different tissues was detected to evaluate whether the tissues had cancer tissue invasion.

SUMMARY:
Accurate evaluation of tumor boundaries in breast-conserving surgery is closely associated with reducing the second operation of patients. Meanwhile, accurately assessing sentinel lymph node (SLN) metastasis is crucial for determining the extent of axillary lymph node dissection (ALND) and minimizing complications. Near-infrared-II (NIR-II) fluorescence imaging using molecular agents has shown promise for in situ imaging during resection. However, very effective probes can be applied to clinical trials up to now, which limits the clinical application of fluorescence imaging. Here we developed a new technology that can quickly differentiation between cancer and para-cancer tissue as well as metastatic and normal sentinel lymph nodes(SLN). In brief, the fresh tissues were incubated with the probe immediately after intraoperative resection and imaged to identify the tumor area and distinguish the metastatic status of SLN. The accuracy of fluorescence imaging was confirmed by pathological diagnosis.

DETAILED DESCRIPTION:
After enrollment, the patients received surgical treatment according to clinical diagnosis and treatment.During the operation, the excised breast tissue and SLN was incubated, and the specific procedure was as follows.

1. Preparation of the incubation solution: The probe was dissolved in phosphate buffer saline(PBS) buffer as the incubation solution at room temperature in the dark,with varying concentrations (12.5, 25, 50,100 ug/mL).
2. In vitro incubation of fresh breast cancer or SLN tissues: The fresh excision breast cancer and SLN tissues were completely soaked in the incubation solution for about 1,3, 5, 7 or 10 minutes, followed by 5 minutes rinse with PBST buffer (PBS with Tween 20) and drying with the use of absorbent paper.
3. Analysis of the images in the "Digital Precision Medicine(DPM)" NIR-II system. The DPM parameter was set up before scaling. Then fluorescence imaging was performed with the DPM NIR-II system. And the result was analyzed to identify the tumor area and distinguish the metastatic status of SLN.
4. Confirmed the diagnosis by pathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-75 years of age
* Female
* Patients presenting with a breast nodule or mass presumed to be resectable on pre-operative assessment
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Patients unable to participate in the consent process
* Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc
* Other conditions that the researcher considers inappropriate to participate in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 40 female patients, aged 18 to 75 years, who have been assessed to have resectable breast nodules or masses and are scheduled to undergo surgery. During the surgery, the resected tumors and lymph nodes will be incubated with theNIR-II probe(ICG-POL6326) solution, and NIR-II fluorescence signals from the tissues will be collected.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Expression of the CXCR4 in the tumor | 2 year
  Ability of the imaging system to detect the expression of the CXCR4 in the mass (i.e tumor).
Uptake of the dye by the tissue(i.e tumor,metastatic SLN) | 2 year
  Ability of the imaging system to discern the uptake of the dye by the tumor or metastatic SLN . Detected with imaging probe.
False positive rates of the NIR-II probe (ICG-POL6326) | 2 year
  Microscopic examination and immunohistochemistry of tumor performed by a pathologist. This will allow investigators to compare pathology results with fluorescence images taken by imaging probe to calculate false positive (i.e., identification of non CXCR4-positive tumors) rates of ICG-POL6326.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39413161/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37540231/